CLINICAL TRIAL: NCT04002908
Title: Low-birthweight Infant Feeding Exploration
Acronym: LIFE
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Emory University (Other); Boston Children's Hospital (Other); Brigham and Women's Hospital (Other); PATH (Other); University of North Carolina, Chapel Hill (Other); Jawaharlal Nehru Medical College (Other); Muhimbili University of Health and Allied Sciences (Other); University of North Carolina (Other); Ariadne Labs (Other)
Responsible Party: Principal Investigator, Katherine Semrau, Director of BetterBirth Program at Ariadne Labs; Assistant Professor, Harvard School of Public Health (HSPH)
Other Study IDs: HSPH OPP1192260
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Low Birthweight; Pre-Term
Keywords: Infant Health; Low and Middle Income Countries [LMIC]; Maternal Health; Infant Feeding; Low Birthweight
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- In-facility Observations: Mothers and their LBW babies will be observed starting within 6 hours of birth until the baby is discharged from the health facility.
- Prospective cohort study - Quantitative: Mothers and their low-birth weight babies will be enrolled 72 hours after birth and followed through 12 months postpartum. The prospective cohort survey (which includes anthropometric measurements and feeding observations) occurs at multiple time points over this 12-month period.
- Prospective cohort study - Qualitative: Research specialists at each site will be speaking to key informants (includes doctors, nurses, midwives, community health workers (CHWs), Ministry of Health (MOH) officials, supply chain & milk bank experts) who are knowledgeable about breastfeeding policy, supply chain, or milk banks. Clinicians in study health facilities who work on labor and delivery, postnatal, newborn and neonatal ICU wards. They participate in In-depth interviews. Mothers, family members and health care workers of LBW babies, as well as community leaders (including religious leaders) who are knowledgeable about infant feeding in their communities will participate in focus group discussions. Focus group discussion will take up to 2 hours. In-depth interviews will take up to 1 hour.
  Mothers (6-month extension): Mothers chosen and consented for in-depth interviews (IDIs) will include those currently enrolled in the prospective cohort. Additionally, their infants need to be between 9 and 12 months of age.
- Retrospective Chart review: The retrospective chart review is a review of secondary data of mothers and their LBW babies who were born in the study health facilities prior to the start of the study.
- Donor Human Milk Readiness Assessment: Key stakeholders in the area of newborn health who determine policy and procedures or who are directly involved with the provision of care. This includes clinicians, nurses, lactation/nutrition specialists, hospital leadership and/or Ministry of Health officials present in the study health facilities.
  This is a one-time data collection exercise in the form of either: (1) a largely qualitative facility readiness assessment tool with some qualitative questions for facility staff or (2) a facility tool observing the "flow of milk" along with key informant interviews in the study facilities. This could take anywhere from 1hr to a day depending on the tool administered, key informants involved and size of the study facility.

SUMMARY:
Globally, 15% of all babies, amounting to 20 million infants each year, are born low birthweight (LBW), defined less than 2500 grams (5.5 lbs). Compared to normal weight infants, LBW infants are at higher risk of morbidity, mortality, and poor growth (Risnes et al 2011; Larroque et al 2001; WHO 2006). The main causes of LBW are preterm birth, intrauterine growth restriction (IUGR), or their combination. Unfortunately, there is a paucity of information around feeding practices and optimal feeding strategies for this population, particularly for LBW infants who struggle with breastfeeding or growth. This study hopes to address these gaps.

DETAILED DESCRIPTION:
The Low-birthweight Infant Feeding Exploration (LIFE)(original grant 0-6 months of age) and the 6- month extension (6-12 months of age) will fill a critical data gap in the field of newborn care regarding vulnerability and feeding of LBW infants. The investigators aim to establish the background information required to set up and test the most efficient and feasible infant feeding strategies for LBW infants: first to support breastfeeding, and then to support infants who are nutritionally at risk in the first 6 month of life in low and middle income countries (LMIC). The investigators will explore all three infant feeding options currently included in the WHO guidelines for LBW infants (WHO 2011), namely mother's own milk (MOM), donor human milk (DHM), and breast milk substitute or formula (BMS), in that order. This work will provide much-needed evidence to inform infant feeding guidelines.

In addition, this 6-month extension will allow for a more comprehensive exploration and understanding of feeding options for LBW infants from 6 to 12 months of age, accounting for timing of introduction of complementary liquids and foods, changes in feeding types, growth and health outcomes over the entire infancy period. This will contribute significantly and allow for high quality data to describe the burden of disease across sites. Specifically, we will be able to describe the following for LBW infants:

* Growth trajectories from 0 to 12 months of age
* Patterns and timing of complementary feeding and continued breastfeeding/breastmilk consumption
* Common infant morbidities and timing of mortality
* Maternal demographics, well-being and environmental factors affecting infant feeding and growth

The overall study goal is to understand feeding options for LBW infants in LMIC settings, including current feeding practices, health outcomes, and potential interventions. The study will take place in four study sites located in three countries: Tanzania, Malawi, and India. Each study site will encompass 2 to 5 individual study facilities. The three study objectives under the goal include:

1. Understand the current practices and standard of care (SOC) for feeding LBW infants
2. Define and document the key outcomes (including growth, morbidity, and lack of success on MOM) for LBW infants under current practices
3. Assess the acceptability and feasibility of a system-level IYCF intervention and the proposed infant feeding options for LBW infants

The investigators will also use the results of this work to design ways to support exclusive breastfeeding (including strategies for feeding with MOM), and to support other options, when mother's own milk (MOM) is unavailable or infants are nutritionally at risk. To do this, the investigators will engage in discussion and consensus-building activities among study staff and key stakeholders, using the collected study data to inform feasible, acceptable Infant and Young Child Feeding (IYCF) strategies for LBW infants that include specific options for those who are nutritionally at risk. The strategies will be tailored to the country as much as possible. A primary product for this later stage will be a white paper documenting key findings from the research and proposing feeding strategies for LBW infants in study sites.

ELIGIBILITY:
Inclusion Criteria:

* Infant birthweight between 1500 and <2500g (according to chart and then verified by study staff).
* Residence within catchment area of facility.
* Mother's consent obtained for herself and infant.
* Newborns must be enrolled within 72 hours of birth.
* Women (mothers) who are of age of majority in their respective countries.

Exclusion Criteria:

* Mother does not meet the local age of majority.
* Infant very low birthweight <1500g.
* Infant has congenital abnormality that interferes with feeding, which includes: Cleft lip or palate; Hydrocephalus; Gastrointestinal tract anomalies including gastroschisis, omphalocele, or anal atresia; Neural tube defects; Congenital cardiac defects; Suspected Trisomy 21; Suspected TORCH infection such as congenital rubella, cytomegalovirus (CMV), toxoplasmosis, or syphilis.
* Critical or severe illness jeopardizing early survival, specifically, investigators will exclude infants with severe encephalopathy as determined by modified Sarnat criteria.
* If the Infant dies before enrollment can occur.
* Infant has a twin or triplet that has died.
* Plans to leave the study area before end of data collection.
* Infants must be enrolled in the prospective study within 72 hours of birth. If the infant is older than 72 hours at the time of screening, s/he will be ineligible for the study.
* Maternal death: The study will exclude cases of maternal death that occur during labor and delivery (or at any time before the consenting process would begin for this study).
* Maternal deaths will count as an exclusion criterion for the prospective cohort if they occur before enrollment. In the event that a mother dies at any time after enrollment the infant will still be retained in the cohort.

  6-Month Extension Study Criteria:

Inclusion criteria for the mother/infant pair are:

* Currently enrolled in the LIFE study and fulfills all original inclusion criteria.
* Mother's or surrogate consent obtained for herself and infant for another 6 months of follow up.

Exclusion criteria for the mother/infant pair are:

• Not previously enrolled in the LIFE study in addition to all original exclusion criteria.

Ages: 16 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Mothers and their LBW babies who are either born in the study health facilities or arrive within 72 hours of birth and meet eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 3188 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Semrau, PhD, MPH, Principal Investigator — Ariadne Labs
Locations (3):
- Jawaharlal Nehru Medical College, Belagavi, India
- UNC Project Malawi (UNCPM), Lilongwe, Malawi
- Muhas/ Hsph, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset will be available through Harvard Dataverse for the LIFE data. A prospective cohort data set will be available and a in-facility observation cohort will be available.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available 12 months after study completion and available indefinitely.
Access Criteria: Those who wish to use the dataset must register for access through Harvard Dataverse. There are no fees or charges associated with data access.
URL: https://dataverse.harvard.edu/dataverse/BetterBirthData

REFERENCES:
- [Derived] Mvalo T, Dhaded SM, Manji KP, Vesel L, Semrau KEA, Kisenge R, Somji S, Chiume M, Saidi F, Hoffman IF, Vernekar S, Bellad R, Koppad B, Tuller DE, Mokhtar R, Lee ACC, North K, Sudfeld CR. Mortality, morbidity and growth among moderately low birthweight infants in India, Malawi, and Tanzania. BMC Pediatr. 2025 Apr 23;25(1):316. doi: 10.1186/s12887-025-05668-8. PMID 40264138
- [Derived] Vesel L, Bellad RM, Manji K, Saidi F, Velasquez E, Sudfeld CR, Miller K, Bakari M, Lugangira K, Kisenge R, Salim N, Somji S, Hoffman I, Msimuko K, Mvalo T, Nyirenda F, Phiri M, Das L, Dhaded S, Goudar SS, Herekar V, Kumar Y, Koujalagi MB, Guruprasad G, Panda S, Shamanur LG, Somannavar M, Vernekar SS, Misra S, Adair L, Bell G, Caruso BA, Duggan C, Fleming K, Israel-Ballard K, Fishman E, Lee ACC, Lipsitz S, Mansen KL, Martin SL, Mokhtar RR, North K, Pote A, Spigel L, Tuller DE, Young M, Semrau KEA; LIFE study team. Feeding practices and growth patterns of moderately low birthweight infants in resource-limited settings: results from a multisite, longitudinal observational study. BMJ Open. 2023 Feb 15;13(2):e067316. doi: 10.1136/bmjopen-2022-067316. PMID 36792338
- [Derived] Vesel L, Spigel L, Behera JN, Bellad RM, Das L, Dhaded S, Goudar SS, Guruprasad G, Misra S, Panda S, Shamanur LG, Vernekar SS, Hoffman IF, Mvalo T, Phiri M, Saidi F, Kisenge R, Manji K, Salim N, Somji S, Sudfeld CR, Adair L, Caruso BA, Duggan C, Israel-Ballard K, Lee AC, Martin SL, Mansen KL, North K, Young M, Benotti E, Marx Delaney M, Fishman E, Fleming K, Henrich N, Miller K, Subramanian L, Tuller DE, Semrau KE. Mixed-methods, descriptive and observational cohort study examining feeding and growth patterns among low birthweight infants in India, Malawi and Tanzania: the LIFE study protocol. BMJ Open. 2021 Dec 2;11(12):e048216. doi: 10.1136/bmjopen-2020-048216. PMID 34857554
- See also: Harvard Dataverse with LIFE study data available. — https://dataverse.harvard.edu/dataverse/BetterBirthData

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The LIFE study did not involve an intervention. Enrollment of the prospective cohort was of mother-infant dyads; we have reported baseline data of the respective individuals. Outcome measurement is at the infant level. Similarly, for the in-facility observation cohort, we have reported baseline characteristics of individuals (mothers and infants); however, the outcomes are focused on infants. Thus, we have reported outcomes at that level.
Units Other Than Participants: facilities
Groups:
- In-facility Observations: Moderately low birthweight infants (1500 to <2500g) and their mothers (i.e. dyads) were enrolled for observation while in the post-natal ward or neonatal intensive care unit.
- Prospective Cohort Study - Qualitative: Qualitative interviews: Focus Group Discussions (FGDs) were conducted with mothers, family members, and community leaders; In-depth interviews (IDIs) were completed with Health care providers, government officials, and supply chain and donor human milk experts
- LIFE Study: Retrospective Chart Review & Donor Human Milk Readiness Assessment: Medical records of moderately low birthweight infants from 12 months before study initiation were reviewed from facilities involved in the LIFE study. Additionally, a Donor Human Milk Readiness Assessment was conducted at each of the participating facilities.
Period: Overall Study
Arm/Group | Prospective Cohort Study - Quantitative | In-facility Observations | Prospective Cohort Study - Qualitative | LIFE Study: Retrospective Chart Review & Donor Human Milk Readiness Assessment
Started | 2184; 12 facilities | 290; 12 facilities | 355; 12 facilities | 359; 12 facilities
Completed | 1925; 12 facilities | 290; 12 facilities | 355; 12 facilities | 359; 12 facilities
Not Completed | 259; 0 facilities | 0; 0 facilities | 0; 0 facilities | 0; 0 facilities
Not completed — Death | 41 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 112 | 0 | 0 | 0
Not completed — Lost to Follow-up | 72 | 0 | 0 | 0
Not completed — Infant died, so mother withdrawn | 34 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total 2184 mothers and infants were enrolled in the prospective cohort study (1070 mothers, 1114 infants). For in-facility observation, a separate 290 individuals (142 mothers, 148 infants) were enrolled. Denominators vary by baseline characteristic below. The other 3 cohorts did not have baseline data collected.
Groups:
- In-facility Observations: Moderately low birthweight (1500 to < 2500g) infants and their mothers were enrolled during their admission to the postnatal ward or neonatal intensive care unit.
- Total: Total of all reporting groups
Arm/Group | Prospective Cohort Study - Quantitative | In-facility Observations | Total
Number analyzed (Participants) | 2184 | 290 | 2474
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The numbers shown here are the number of mothers (not the number of infants).Infant age was not collected as all infants were enrolled around the time of birth.
  Years
    number analyzed (Participants) | 1070 | 142 | 1212
    (all) | 25.4 (5.3) | 26.5 (6.1) | 25.8 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We have differentiated the baseline sex between infants and mothers and presented a row for each sub-group
  Participants
    Infant Sex: number analyzed (Participants) | 1114 | 148 | 1262
    Infant Sex: Female | 608 | 85 | 693
    Infant Sex: Male | 506 | 63 | 569
    Mothers sex: number analyzed (Participants) | 1070 | 142 | 1212
    Mothers sex: Female | 1070 | 142 | 1212
    Mothers sex: Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: This is the number of infants and mothers; we have presented data by sub-group.
  Participants
    South Asian Infants: number analyzed (Participants) | 1114 | 148 | 1262
    South Asian Infants | 506 | 73 | 579
    African Infants: number analyzed (Participants) | 1114 | 148 | 1262
    African Infants | 608 | 75 | 683
    South Asian Mothers: number analyzed (Participants) | 1070 | 142 | 1212
    South Asian Mothers | 497 | 72 | 569
    African Mothers: number analyzed (Participants) | 1070 | 142 | 1212
    African Mothers | 573 | 70 | 643
Region of Enrollment [Count of Participants; unit: Participants] — Population: Infants and mothers are presented separately.
  Participants
    Malawi: number analyzed (Participants) | 573 | 70 | 643
    Malawi: Mothers | 273 | 35 | 308
    Malawi: Infants | 300 | 35 | 335
    Tanzania: number analyzed (Participants) | 608 | 75 | 683
    Tanzania: Mothers | 300 | 35 | 335
    Tanzania: Infants | 308 | 40 | 348
    India: number analyzed (Participants) | 1003 | 145 | 1148
    India: Mothers | 497 | 72 | 569
    India: Infants | 506 | 73 | 579
Maternal Education [Count of Participants; unit: Participants] — Population: This is the number of mothers (not the number of infants).
  Participants
    number analyzed (Participants) | 1070 | 142 | 1212
    Primary or less | 501 | 63 | 564
    Secondary or more | 569 | 79 | 648

OUTCOME MEASURES:

1. Primary Outcome: Length-for-Age Z-score
Description: A Child's length-for-age z-score at 6 months of age. Length-for-age z-scores (LAZ) are based on World Health Organization (WHO) child growth standards for term infants and INTERGROWTH-21st standards were used for preterm infants. A LAZ Z-score of 0 represents the population mean and scores below 0 represent a worse outcome. Further, Z-scores less than -2.0 indicates stunting in the infant.
Time Frame: At 6 month of age
Population: Low birth weight infants. This outcome was only collected on the quantitative prospective cohort population.
Measure: Mean (Standard Deviation); unit: Z-score
Groups:
- Prospective Cohort Study - Quantitative: Mothers and their low-birth weight babies will be enrolled 72 hours after birth and followed through 12 months postpartum. The prospective cohort survey (which includes anthropometric measurements and feeding observations) occurs at multiple time points over this 12-month period.
  This outcome (like all others reported) was only assessed in the prospective cohort and not in the in-facility observations, Donor human milk readiness assessment, prospective cohort qualitative or the retrospective chart review.
Arm/Group | Prospective Cohort Study - Quantitative
Number analyzed (Participants) | 1114
Z-score | -1.43 (1.28)

2. Secondary Outcome: Incidence of Diarrheal Disease
Description: Maternal Report of Ever having Diarrheal Disease from weeks 1 to 6 months of age
Time Frame: 6 month postpartum
Population: Low Birth Weight Infants; This outcome was only collected on the quantitative prospective cohort population.
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Cohort Study - Quantitative
Number analyzed (Participants) | 1114
Participants | 130

3. Other Pre Specified Outcome: Weight-for-age Z-score
Description: Child's weight-for-age z-score. Weight-for-age (WAZ) z-scores at 6 months of age were based on WHO growth standards for term infants and INTERGROWTH- 21st standards, for preterm infants. A Z-score of 0 represents the population mean, and Z-scores below 0 represent a worse outcome. Further, WAZ Z-scores less than -2 indicates an infant who is underweight.
Time Frame: At 6 month of age
Population: Low Birth Weight Infants; This outcome was only collected on the quantitative prospective cohort population.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Prospective Cohort Study - Quantitative
Number analyzed (Participants) | 1114
Z-score | -1.23 (1.20)

4. Other Pre Specified Outcome: Percentage of Infants Malnourished at 6 Months
Description: Infants who were stunted and/or wasted and/or underweight according to WHO Growth Standards at 6 months of age. A Z-score of 0 represents the population mean, and Z-scores below 0 represent a worse outcome Infants who have Z-score (weight for age; length for age; or weight for length) less than -2 are considered malnourished.
Time Frame: 6 months of age
Population: Low birth weight infants; This outcome was only collected on the quantitative prospective cohort population.
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Cohort Study - Quantitative
Number analyzed (Participants) | 1114
Participants | 373

5. Other Pre Specified Outcome: Percentage of Infants Malnourished at 12 Months
Description: Infants who were stunted and/or wasted and/or underweight according to WHO Growth Standards at 12 months of age. A Z-score of 0 represents the population mean, and Z-scores below 0 represent a worse outcome Infants who have Z-score (weight for age; length for age; or weight for length) less than -2 are considered malnourished.
Time Frame: 12 months of age
Population: Low birth weight infants
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Cohort Study - Quantitative
Number analyzed (Participants) | 1114
Participants | 518

6. Other Pre Specified Outcome: Weight-for-age Z-score
Description: Child's weight-for-age z-score. Child's weight-for-age z-score. Weight-for-age (WAZ) z-scores at 12 months were based on WHO growth standards for term infants and preterm infants. A Z-score of 0 represents the population mean, and Z-scores below 0 represent a worse outcome. Further, WAZ Z-scores less than -2 indicates an infant who is underweight.
Time Frame: At 12 month of age
Population: Low Birth Weight Infants; This outcome was only collected on the quantitative prospective cohort population.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Prospective Cohort Study - Quantitative
Number analyzed (Participants) | 1114
Z-score | -1.28 (1.12)

7. Primary Outcome: Length-for-Age Z-score
Description: A Child's length-for-age z-score at 12 months of age. A Child's length-for-age z-score at 12 months of age. Length-for-age (LAZ) z-scores were based on World Health Organization (WHO) growth standards for term infants and preterm infants; we corrected for gestational age (GA) for preterm infants. A LAZ z-score of 0 represents the population mean and scores below 0 represent a worse outcome. Further, Z-scores less than -2.0 indicates an infant who is underweight.
Time Frame: At 12 month of age
Population: Low birth weight infants; This outcome was only collected on the quantitative prospective cohort population.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Prospective Cohort Study - Quantitative
Number analyzed (Participants) | 1114
Z-score | -1.58 (1.21)

ADVERSE EVENTS:
Time Frame: 1 year
Description: All-cause mortality was collected from prospective cohort mothers, infants, and infants in the in-facility cohort. Adverse events (AE) were only collected on infants and mothers in prospective cohorts and in-facility cohort: infants. AE was monitored so that specific AE Terms could not be separated for infants (n=1114). We did not collect AE data on the qualitative cohorts (mothers or infants) or the retrospective chart review/donor human milk readiness assessment.
Groups:
- Prospective Cohort Study - Quantitative: Infants; Prospective Cohort Study - Quantitative: Mothers: Mothers and their low-birth weight babies will be enrolled 72 hours after birth and followed through 12 months postpartum. The prospective cohort survey (which includes anthropometric measurements and feeding observations) occurs at multiple time points over this 12-month period.
  Only the prospective cohort quantitative arm is included in adverse arm reporting since this was the longitudinal, prospective cohort for which we reported outcomes and reported adverse events.
- In-facility Observations: Low-birthweight infants were followed during their in-facility stay and followed until facility discharge.
Arm/Group | Prospective Cohort Study - Quantitative: Infants | Prospective Cohort Study - Quantitative: Mothers | In-facility Observations
All-Cause Mortality (participants affected / at risk) | 37/1114 | 4/1070 | 3/142
Serious Adverse Events (participants affected / at risk) | 172/1114 | 22/1070 | 8/142
Other Adverse Events (participants affected / at risk) | 0/1114 | 0/1070 | 0/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prospective Cohort Study - Quantitative: Infants (N=1114) | Prospective Cohort Study - Quantitative: Mothers (N=1070) | In-facility Observations (N=142)
Malnutrition (Gastrointestinal disorders) | 113 | 10 | 0
Severe Illness (General disorders) | 7 | 0 | 0
Other Illness (General disorders) | 50 | 12 | 8
Unknown Illness (General disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT04002908/Prot_SAP_001.pdf
  • Informed Consent Form (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT04002908/ICF_002.pdf